CLINICAL TRIAL: NCT07053553
Title: Determining the Effect of Home Care Training on Anxiety and Depression Levels of Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hatun Erkuran, Lecturer, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Gumushane University
Record Dates: First submitted 2025-06-18; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Being Registered With Kelkit District State Hospital Home Health Unit; Being a Home Care Patient
Keywords: Caregivers; Health Education; Home Care; Home Nursing; Mental Health
MeSH Terms: conditions — Health Education; Psychological Well-Being | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (n=21) (Experimental): Experimental (n=21)
  Interventions: Other: Education
- control groups (No Intervention): control (n=21) groups

INTERVENTIONS:
Other: Education — It was planned to provide bed bath training to inpatients because 90.5% of the caregivers of the patients in the experimental group wanted to receive bed bath training.
  Arms: Experimental (n=21)

SUMMARY:
This study was conducted to determine the effects of home care training given to caregivers of patients receiving home care services on the anxiety and depression levels of the caregivers. The study was conducted as a pre-test/post-test, randomized controlled quasi-experimental with a total of 42 patients and caregivers receiving home care services, 21 in the experimental group and 21 in the control group, registered at the Home Health Unit of Kelkit District State Hospital in Gümüşhane province between September 2023 and December 2024. Caregiver Information Form, Beck Anxiety Inventory, Beck Depression Inventory, and Patient Body Bath Caregiver Follow-up Form were used as data collection tools. The caregivers in the experimental group were asked about which subject they wanted to receive training, and it was determined that they wanted to receive training on in-bed body bath, and patient body bath caregiver training was planned and implemented. No application was made to the caregivers in the control group. SPSS 22 statistical program was used in the analysis of the data and the significance level was accepted as p<0.05.

DETAILED DESCRIPTION:
The research was conducted in the homes of patients and caregivers who were registered with the Home Health Unit of Kelkit District State Hospital in Gümüşhane province and received home care services. Data collection tools were created between May and August 2023. Research data were collected between September 2023 and December 2024. The research was completed by data analysis and reporting between January and March 2025. The caregivers included in the research sample were listed consecutively according to the order of their application to the Home Health Unit of Kelkit District State Hospital in Gümüşhane province and were divided into experimental (n=23) and control (n=22) groups via the internet using the simple random sampling method. After 3 caregivers did not want to participate in the study, a study was conducted with 42 caregivers (21 experimental, 21 control). The first interview with the experimental (n=21) and control (n=21) groups was conducted face to face at the caregivers' homes, and a pre-test was conducted after the written consent form was obtained from the caregivers who agreed to participate in the study. In the pre-test application, the BVBF, Beck Anxiety Inventory, and Beck Depression Inventory were filled out. A second interview was conducted to determine the issues that the caregivers in the experimental group had difficulty with, experienced stress, felt the need for training, and wanted to receive training during care practices, and it was found that the majority of the caregivers wanted to receive patient bed bath training.After the second interview, bed bath training was planned for the caregivers of the patients in the experimental group, the training content and patient body bath caregiver follow-up forms were created, and the created training plan was sent for expert opinion in terms of suitability. After the expert opinion was received, a third interview was planned with the caregivers of the patients in the experimental group, during the interview, the caregivers were asked to apply body bath to the patient, the caregiver was observed while applying body bath to the patient, and in order to evaluate the incomplete/faulty practices of the caregiver during the application, the HVBBVİF was filled in by the researcher while the caregiver was performing the application.

1 week after the third interview, the 4th interview was conducted with the caregivers of the patients in the experimental group, and the bed bath training was demonstrated and applied by the researcher to the patient's caregiver. 1 week after the fourth interview, the 5th interview was conducted with the caregivers of the patients in the experimental group, and the HVBBVİF was filled in by the researcher while the caregiver was performing body bath to the patient, and the incomplete/faulty practices were corrected by the researcher with immediate feedback. Two weeks after the 5th interview, the 6th interview was conducted with the caregivers of the patients in the experimental group, the caregiver applied the bed bath to the patient, and the HVBBVİF was filled in by the researcher. One week after the sixth interview, the 7th interview was conducted with the experimental and control groups, and for the post-test application, the "BVBF", "Beck Anxiety Inventory", and "Beck Depression Inventory" were filled in again.

ELIGIBILITY:
Inclusion Criteria:

* Being registered with the Kelkit District State Hospital Home Health Unit
* Being willing to participate in the research
* Being able to read and write in Turkish and be able to communicate
* Not having vision or hearing loss
* Being able to make phone calls

Exclusion Criteria:

* Not registered with Kelkit District State Hospital Home Health Unit
* Not volunteering to participate in the research
* Not knowing how to read and write in Turkish and not being able to communicate
* Having vision and hearing loss
* Not being able to communicate by phone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Home care training has an effect on anxiety and depression levels of caregivers. | from registration to the end of the 12th week
  Beck Anxiety Inventory is a self-assessment scale. It is a Likert-type scale consisting of 21 items. According to the scale score ranges, 0-7 points indicate minimal anxiety, 8-15 points indicate mild anxiety, 16-25 points indicate moderate anxiety, and 26-63 points indicate severe anxiety. The Beck Depression Inventory was developed by Beck in 1961 to measure the risk of depression in adults, the level of depressive symptoms, and the change in severity. The scale consists of 21 items. It is a four-degree self-assessment scale. The highest score that can be obtained from the scale is 63. The cut-off score was accepted as 17. According to the scale score ranges, 0-9 points indicate minimal depressive symptoms, 10-16 points indicate mild depressive symptoms, 17-29 points indicate moderate depressive symptoms, and 30 and above points indicate severe depressive symptoms.
Home care training has an impact on hospital admissions of patients receiving home care services. | from registration to the end of the 12th week
  It is aimed to reduce the frequency of patients' hospital admissions after home care training.

SECONDARY OUTCOMES:
Home care training has an impact on the frequency of home care patients applying to the home care unit. | from registration to the end of the 12th week
  It is aimed to reduce the frequency of patients applying to home care units after home care training.

CONTACTS AND LOCATIONS:
Overall Officials: Havva Karadeniz, Assist.Prof.PhD, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gümüşhane University, Gümüşhane, Gümüşhane Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: SAP, ICF, CSR
Time Frame: September 2024- July 2025

REFERENCES:
- See also: Beck Anxiety — https://www.scribd.com/document/715100262/Turkish-Version-of-the-Beck-Anxiety-Inventory-Psychometric-Properties
- See also: Beck Depression scales — https://psikolog.org.tr/tr/yayinlar/dergiler/1031828/tpd1300443319890000m000366.pdf